CLINICAL TRIAL: NCT01054456
Title: A Multicenter, Open-Label, Single-Arm Evaluation of Palonosetron for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) in Subjects Who Have Experienced CINV(Chemotherapy-Induced Nausea and Vomiting) During the Previous Cycle of Low Emetogenic Chemotherapy (LEC)
Brief Title: A Study of Palonosetron for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) in Participants Who Have Experienced CINV(Chemotherapy-Induced Nausea and Vomiting) During the Previous Cycle of Low Emetogenic Chemotherapy (LEC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PALO-08-13
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2011-01

CONDITIONS: Patients With Confirmed Malignant Disease to Receive Low Emetogenic Chemotherapy (LEC) or Who Experienced at Least Nausea and Vomiting During Last Cycle of LEC
Keywords: LEC; Low Emetogenic Chemotherapy; Nausea and Vomiting; Nausea; Vomiting; Anti- emetic
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants: Palonosetron 0.25 mg/5 mL (Experimental): Participants will receive palonosetron 0.25 milligram (mg) per (/) 5 milliliter (mL) intravenous injection 30 minutes prior to receiving a low emetogenic chemotherapy (LEC) agent on Day 1.
  Interventions: Drug: palonesetron

INTERVENTIONS:
Drug: palonesetron — One dose administered intravenously 30 minutes pre-chemotherapy

SUMMARY:
This study is designed to assess the safety and efficacy of palonesetron in preventing chemotherapy-induced nausea and vomiting (CINV) when administered to participants who have experienced either vomiting and or at least moderate nausea during their last cycle of low emetogenic chemotherapy.

DETAILED DESCRIPTION:
Palonosetron is currently approved for prevention of acute and delayed nausea and vomiting associated with initial and repeat CINV caused by moderate and highly emetogenic chemotherapy. This study is designed to assess the safety and efficacy of palonesetron in preventing CINV when administered to patients who have experienced either vomiting and or at least moderate nausea during their last cycle of low emetogenic chemotherapy.

Palonosetron will be given intravenously approximately 30 minutes prior to the start of the chemotherapy regimen. Efficacy and safety including episodes of nausea, retching and or vomiting will be assessed over five 24 hour periods starting on Day 1 and ending on Day 6 in patient diaries. On Day 2 and Day 6 a FLIE (Functional Living Index- Emesis) assessment will also be completed in order to help evaluate the patient's quality of life from the start of the chemotherapy cycle through Day 6.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible for enrollment, subjects must meet the following inclusion criteria:

1. Provide written informed consent
2. Male or female ≥18 years of age
3. Histologically or cytologically confirmed malignant disease
4. Karnofsky Index of 50%
5. Experienced either vomiting and/or at least moderate nausea during their last cycle of LEC
6. Scheduled to receive, on Study Day 1, a single dose of one of the qualifying LEC agents listed in the protocol.
7. Known mild to moderate hepatic, renal or cardiovascular impairment may be enrolled at the discretion of the Investigator Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Inability or unwillingness to understand or cooperate with the study procedures as determined by the Investigator
2. Women who are pregnant, nursing or planning to become pregnant, women of childbearing potential who are not using an effective method of pregnancy prevention (including implants, injectables, combined oral contraceptives, some intrauterine devices, vasectomized partner or sexual abstinence), or women who have had a positive serum pregnancy test at screening or within 7 days prior to receiving chemo on Day 1. Non-childbearing potential includes women who are post-menopausal (12 months of amenorrhea with no other demonstrable cause, in the appropriate age group) or documented surgical sterilization, or hysterectomy at least 3 months before study start.
3. Previous use of palonosetron in association with a LEC regimen
4. Received more than one antiemetic agent for prevention of CINV (Chemotherapy-Induced Nausea and Vomiting) during their last cycle of LEC (other than dexamethasone or prednisone as outlined in number 7 below). The use of an antiemetic in addition to a corticosteroid during the last cycle of LEC is allowed if the corticosteroid is intended for the prophylactic treatment of taxane-related hypersensitivity or pemetrexed-related skin reactions as long as the corticosteroid regimen remains unchanged during the trial
5. Suspected or confirmed ongoing vomiting for any organic etiology (e.g., food poisoning, gastroenteritis, etc)
6. Received any drug with potential anti-emetic effect within 24 hours prior to the start of qualifying LEC agent
7. Scheduled to receive an antiemetic (with the exception of administration of the palonosetron) at any time during the trial, listed below

   -5-HT3 receptor antagonists
   * NK1 receptor antagonists
   * Dopamine receptor antagonists (metoclopramide)
   * Phenothiazine anti-emetics (prochlorperazine, promethazine, thiethylperazine and perphenazine)
   * Diphenhydramine, scopolamine, chlorpheniramine maleate, trimethobenzamide. Diphenhydramine will be allowed if given for prophylactic treatment of hypersensitivity reactions associated with the administration of taxanes (e.g., paclitaxel, docetaxel) and ixabepilone
   * All benzodiazepines except Triazolam or Zolpidem used once at night time due to sleep disturbances
   * Atypical antipsychotic agents with compazine-like activity (e.g., olanzapine, risperidone)
   * Butyrophenones (haloperidol, droperidol)
   * Cannabinoides (tetrahydrocannabinol or nabilone)
   * Any systemic corticosteroid (hydrocortisone, methylprednisolone, prednisone), with the exception of topical or inhaled preparations. Dexamethasone will be allowed if given for prophylactic treatment of hypersensitivity reactions associated with the administration of taxanes (e.g., paclitaxel, docetaxel) or prevention of rash associated with pemetrexed. Prednisone will be allowed if given for as part of standard regimen with mitoxantrone or docetaxel for prostate cancer.
   * Any non-prescription medication, nutritional supplements, vitamins or herbal-type products known to either possibly cause nausea or vomiting, or used to treat nausea or vomiting
8. Having received any investigational drugs or devices within 30 days before study entry
9. Any vomiting, retching, or National Cancer Institute Common Terminology Criteria for Adverse Events, v.3 (NCI CTCAE) Grade 2 to 4 nausea in the 24 hours preceding chemotherapy
10. History of alcohol or drug abuse
11. Scheduled to receive any other emetogenic chemotherapeutic agents during the study other than those specified in this protocol
12. Any known hypersensitivity/contraindication to 5-HT3 antagonists or study drug excipients
13. Scheduled to receive or have received radiotherapy within 1 week prior to or during the study
14. Any condition that, in the judgment of the Principal Investigator, would make a subject ineligible for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-10-27 (Actual); Primary Completion 2010-12-08 (Actual); Study Completion 2010-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Sheridan Clinical Research, Sunrise, Florida
  - Medical and Surgical Specialists, Galesburg, Illinois
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - Trover Center for Clinical Studies; Merle Mahr Cancer Center, Madisonville, Kentucky
  - Hematology- Oncology Associates of Rockland, PC, Nyack, New York
  - Signal Point Clinical Research, Middletown, Ohio
  - Scott and White Clinic- College Station, College Station, Texas
  - Scott and White Healthcare- Round Rock, Round Rock, Texas
  - Scott and White Memorial Hospital, Temple, Texas

REFERENCES:
- [Derived] Hesketh PJ, Morrow G, Komorowski AW, Ahmed R, Cox D. Efficacy and safety of palonosetron as salvage treatment in the prevention of chemotherapy-induced nausea and vomiting in patients receiving low emetogenic chemotherapy (LEC). Support Care Cancer. 2012 Oct;20(10):2633-7. doi: 10.1007/s00520-012-1527-3. Epub 2012 Jun 24. PMID 22733373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 investigative sites in the United States from 27 October 2009 to 08 December 2010.
Pre-assignment Details: A total of 38 participants were screened, of which 02 were screen failures and 36 participants were enrolled and received the study treatment.
Groups:
- All Participants: Palonosetron 0.25 mg/5 mL: Participants received palonosetron 0.25 milligram (mg) per (/) 5 milliliter (mL) intravenous injection 30 minutes prior to receiving a low emetogenic chemotherapy (LEC) agent on Day 1.
Period: Overall Study
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Started | 36
Completed | 35
Not Completed | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received study medication (palonosetron) and had at least 1 safety assessment after treatment.
Groups:
- All Participants: Palonosetron 0.25 mg/5 mL: Participants received palonosetron 0.25 mg/5 mL intravenous injection 30 minutes prior to receiving a LEC agent on Day 1.
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) During Acute Period (0 to 24 Hours) After Receiving Treatment on Day 1
Description: CR was defined as the participants without any emetic episodes and did not use any rescue medication during acute period (0-24 hours). An emetic episode was defined as 1) one occurrence of vomiting, or 2) a sequence of occurrences in very close succession not relieved by a period of relaxation of at least 1 minute, any number of occurrences of unproductive emesis (retches) in a unique 5-minute period, or 3) an episode of retching of less than 5 minute duration combined with vomiting not relieved by a period of relaxation of at least 1 minute. Participants who completed the diary for a given period and had no emetic episodes and no use of rescue medication were considered to have achieved CR, during the period.
Time Frame: From 0 to 24 hours after receiving treatment on Day 1
Population: The intent-to-treat (ITT) population included all participants who received palonosetron, received at least one dose of the qualifying LEC agents on Day 1, and had at least 1 post-chemotherapy efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants | 88.2 [72.5 to 96.7]

2. Primary Outcome: Percentage of Participants With CR During Delayed Period (24 to 120 Hours) After Receiving Treatment on Day 1
Description: CR was defined as the participants without any emetic episodes and did not use any rescue medication during delayed period (24-120 hours). An emetic episode was defined as 1) one occurrence of vomiting, or 2) a sequence of occurrences in very close succession not relieved by a period of relaxation of at least 1 minute, any number of occurrences of unproductive emesis (retches) in a unique 5-minute period, or 3) an episode of retching of less than 5 minute duration combined with vomiting not relieved by a period of relaxation of at least 1 minute. Participants who completed the diary for a given period and had no emetic episodes and no use of rescue medication were considered to have achieved CR, during the period.
Time Frame: From 24 to 120 hours after receiving treatment on Day 1
Population: The ITT population included all participants who received palonosetron, received at least one dose of the qualifying LEC agents on Day 1, and had at least 1 post-chemotherapy efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants | 67.6 [49.5 to 82.6]

3. Primary Outcome: Percentage of Participants With CR During Overall Period (0 to 120 Hours) After Receiving Treatment on Day 1
Description: CR was defined as the participants without any emetic episodes and did not use any rescue medication during overall period (0-120 hours). An emetic episode was defined as 1) one occurrence of vomiting, or 2) a sequence of occurrences in very close succession not relieved by a period of relaxation of at least 1 minute, any number of occurrences of unproductive emesis (retches) in a unique 5-minute period, or 3) an episode of retching of less than 5 minute duration combined with vomiting not relieved by a period of relaxation of at least 1 minute. Participants who completed the diary for a given period and had no emetic episodes and no use of rescue medication were considered to have achieved CR, during the period.
Time Frame: From 0 to 120 hours after receiving treatment on Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants | 67.6 [49.5 to 82.6]

4. Secondary Outcome: Percentage of Participants With CR at Each 24 Hour Interval After Receiving Treatment on Day 1
Description: CR was defined as the participants without any emetic episodes and did not use any rescue medication. An emetic episode was defined as 1) one occurrence of vomiting, or 2) a sequence of occurrences in very close succession not relieved by a period of relaxation of at least 1 minute, any number of occurrences of unproductive emesis (retches) in a unique 5-minute period, or 3) an episode of retching of less than 5 minute duration combined with vomiting not relieved by a period of relaxation of at least 1 minute. Participants who completed the diary for a given period and had no emetic episodes and no use of rescue medication were considered to have achieved CR, during the period.
Time Frame: From 0 to 24 hours, 24 to 48 hours, 48 to 72 hours, 72 to 96 hours and 96 to 120 hours after receiving treatment on Day 1
Population: ITT population included all participants who received palonosetron, received at least one dose of the qualifying LEC agents on Day 1, and had at least 1 post-chemotherapy efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants
  0 to 24 hours | 88.2 [72.5 to 96.7]
  24 to 48 hours | 79.4 [62.1 to 91.3]
  48 to 72 hours | 85.3 [68.9 to 95.0]
  72 to 96 hours | 85.3 [68.9 to 95.0]
  96 to 120 hours | 82.4 [65.5 to 93.2]

5. Secondary Outcome: Percentage of Participants With CR During 0 to 48, 0 to 72, and 0 to 96 Hours After Receiving Treatment on Day 1
Description: as for outcome 4
Time Frame: From 0 to 48 hours, 0 to 72 hours, and 0 to 96 hours after receiving treatment on Day 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants
  0 to 48 hours | 79.4 [62.1 to 91.3]
  0 to 72 hours | 73.5 [55.6 to 87.1]
  0 to 96 hours | 70.6 [52.5 to 84.9]

6. Secondary Outcome: Percentage of Participants With Complete Control During Acute Period (0 to 24 Hours), Delayed Period (24 to 120 Hours), and Overall Period (0 to 120 Hours) After Receiving Treatment on Day 1
Description: Complete Control was defined as the percentage of participants who had a CR and no more than mild nausea. CR was defined as the participants without any emetic episodes and did not use any rescue medication. An emetic episode was defined as 1) one occurrence of vomiting, or 2) a sequence of occurrences in very close succession not relieved by a period of relaxation of at least 1 minute, any number of occurrences of unproductive emesis (retches) in a unique 5-minute period, or 3) an episode of retching of less than 5 minute duration combined with vomiting not relieved by a period of relaxation of at least 1 minute. Participants who completed the diary for a given period and had no emetic episod es and no use of rescue medication were considered to have CR during the period. Those same participants were considered complete control for the period if they had no more than mild nausea during the period.
Time Frame: From 0 to 24 hours, 24 to 120 hours, and 0 to 120 hours after receiving treatment on Day 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants
  Acute (0 to 24 hours) | 85.3 [68.9 to 95.0]
  Delayed (24 to 120 hours) | 64.7 [46.5 to 80.3]
  Overall (0 to 120 hours) | 64.7 [46.5 to 80.3]

7. Secondary Outcome: Percentage of Participants With Complete Control at Each 24 Hours Interval After Receiving Treatment on Day 1
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants
  0 to 24 hours | 85.3 [68.9 to 95.0]
  24 to 48 hours | 76.5 [58.8 to 89.3]
  48 to 72 hours | 76.5 [58.8 to 89.3]
  72 to 96 hours | 82.4 [65.5 to 93.2]
  96 to 120 hours | 79.4 [62.1 to 91.3]

8. Secondary Outcome: Percentage of Participants With Complete Control During 0 to 48, 0 to 72, and 0 to 96 Hours After Receiving Treatment on Day 1
Description: as for outcome 6
Time Frame: From 0 to 48 hours, 0 to 72 hours, and 0 to 96 hours after receiving treatment on Day 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participant
  0 to 48 hours | 76.5 [58.8 to 89.3]
  0 to 72 hours | 70.6 [52.5 to 84.9]
  0 to 96 hours | 67.6 [49.5 to 82.6]

9. Secondary Outcome: Percentage of Participants With No Emetic Episodes During Acute Period (0 to 24 Hours), Delayed Period (24 to 120 Hours), and Overall Period (0 to 120 Hours) After Receiving Treatment on Day 1
Description: An emetic episode was defined as 1) one occurrence of vomiting, or 2) a sequence of occurrences in very close succession not relieved by a period of relaxation of at least 1 minute, any number of occurrences of unproductive emesis (retches) in a unique 5-minute period, or 3) an episode of retching of less than 5 minute duration combined with vomiting not relieved by a period of relaxation of at least 1 minute.
Time Frame: From 0 to 24 hours, 24 to 120 hours, and 0 to 120 hours after receiving treatment on Day 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants
  Acute (0 to 24 hours) | 91.2 [76.3 to 98.1]
  Delayed (24 to 120 hours) | 79.4 [62.1 to 91.3]
  Overall (0 to 120 hours) | 79.4 [62.1 to 91.3]

10. Secondary Outcome: Percentage of Participants With No Emetic Episodes At Each 24 Hours Interval After Receiving Treatment on Day 1
Description: as for outcome 9
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants
  0 to 24 hours | 91.2 [76.3 to 98.1]
  24 to 48 hours | 94.1 [80.3 to 99.3]
  48 to 72 hours | 88.2 [72.5 to 96.7]
  72 to 96 hours | 91.2 [76.3 to 98.1]
  96 to 120 hours | 88.2 [72.5 to 96.7]

11. Secondary Outcome: Percentage of Participants With No Emetic Episodes During 0 to 48 Hours, 0 to 72 Hours, and 0 to 96 Hours After Receiving Treatment on Day 1
Description: as for outcome 9
Time Frame: From 0 to 48 hours, 0 to 72 hours, and 0 to 96 hours after receiving treatment on Day 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants
  0 to 48 hours | 91.2 [76.3 to 98.1]
  0 to 72 hours | 85.3 [68.9 to 95.0]
  0 to 96 hours | 85.3 [68.9 to 95.0]

12. Secondary Outcome: Percentage of Participants With Nausea Based on Severity and Intensity During Acute Period (0 to 24 Hours), Delayed Period (24 to 120 Hours), and Overall Period (0 to 120 Hours) After Receiving Treatment on Day 1
Description: The 4-point Likert scale was used to measure the severity and intensity of nausea. The participant was asked "How much nausea did you experience on average during the last 24 hours?" The scale was defined as follows: 0 = none, 1 = mild, 2 = moderate, 3 = severe.
Time Frame: From 0 to 24 hours, 24 to 120 hours, and 0 to 120 hours after receiving treatment on Day 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants
  Acute (0 to 24 hours); None | 73.5 [55.6 to 87.1]
  Acute (0 to 24 hours); Mild | 11.8 [3.3 to 27.5]
  Acute (0 to 24 hours); Moderate | 11.8 [3.3 to 27.5]
  Acute (0 to 24 hours); Severe | 2.9 [0.1 to 15.3]
  Delayed (24 to 120 hours), None | 52.9 [35.1 to 70.2]
  Delayed (24 to 120 hours), Mild | 26.5 [12.9 to 44.4]
  Delayed (24 to 120 hours), Moderate | 11.8 [3.3 to 27.5]
  Delayed (24 to 120 hours), Severe | 8.8 [1.9 to 23.7]
  Overall (0 to 120 hours); None | 50.0 [32.4 to 67.6]
  Overall (0 to 120 hours); Mild | 26.5 [12.9 to 44.4]
  Overall (0 to 120 hours); Moderate | 14.7 [5.0 to 31.1]
  Overall (0 to 120 hours); Severe | 8.8 [1.9 to 23.7]

13. Secondary Outcome: Percentage of Participants With Nausea Based on Severity and Intensity At Each 24 Hours Interval After Receiving Treatment on Day 1
Description: as for outcome 12
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants
  0 to 24 hours: None | 73.5 [55.6 to 87.1]
  0 to 24 hours: Mild | 11.8 [3.3 to 27.5]
  0 to 24 hours: Moderate | 11.8 [3.3 to 27.5]
  0 to 24 hours: Severe | 2.9 [0.1 to 15.3]
  24 to 48 hours: None | 73.5 [55.6 to 87.1]
  24 to 48 hours: Mild | 11.8 [3.3 to 27.5]
  24 to 48 hours: Moderate | 11.8 [3.3 to 27.5]
  24 to 48 hours: Severe | 2.9 [0.1 to 15.3]
  48 to 72 hours: None | 76.5 [58.8 to 89.3]
  48 to 72 hours: Mild | 5.9 [0.7 to 19.7]
  48 to 72 hours: Moderate | 11.8 [3.3 to 27.5]
  48 to 72 hours: Severe | 5.9 [0.7 to 19.7]
  72 to 96 hours: None | 67.6 [49.5 to 82.6]
  72 to 96 hours: Mild | 20.6 [8.7 to 37.9]
  72 to 96 hours: Moderate | 8.8 [1.9 to 23.7]
  72 to 96 hours: Severe | 2.9 [0.1 to 15.3]
  96 to 120 hours: None | 82.4 [65.5 to 93.2]
  96 to 120 hours: Mild | 11.8 [3.3 to 27.5]
  96 to 120 hours: Moderate | 5.9 [0.7 to 19.7]
  96 to 120 hours: Severe | 0 [0 to 0]

14. Secondary Outcome: Percentage of Participants With Nausea Based on Severity and Intensity During 0 to 48, 0 to 72, and 0 to 96 Hours After Receiving Treatment on Day 1
Description: as for outcome 12
Time Frame: From 0 to 48 hours, 0 to 72 hours, and 0 to 96 hours after receiving treatment on Day 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
percentage of participants
  0 to 48 hours: None | 67.6 [49.5 to 82.6]
  0 to 48 hours: Mild | 14.7 [5.0 to 31.1]
  0 to 48 hours: Moderate | 11.8 [3.3 to 27.5]
  0 to 48 hours: Severe | 5.9 [0.7 to 19.7]
  0 to 72 hours: None | 61.8 [43.6 to 77.8]
  0 to 72 hours: Mild | 14.7 [5.0 to 31.1]
  0 to 72 hours: Moderate | 14.7 [5.0 to 31.1]
  0 to 72 hours: Severe | 8.8 [1.9 to 23.7]
  0 to 96 hours: None | 52.9 [35.1 to 70.2]
  0 to 96 hours: Mild | 23.5 [10.7 to 41.2]
  0 to 96 hours: Moderate | 14.7 [5.0 to 31.1]
  0 to 96 hours: Severe | 8.8 [1.9 to 23.7]

15. Secondary Outcome: Mean Change From Follow Up Period (Day 2-5) in Scores on Functional Living Index-Emesis [FLIE] Assessment Questionnaires to the End of Study (Day 8)
Description: FLIE is a patient-completed quality of life assessment modified from the original Functional Living Index - Cancer questionnaire. FLIE contains two domains: nausea and vomiting with nine items in each domain. The first item asks the patient to rate how much nausea (or vomiting) has occurred over a 5 day period. The remaining eight items ask patients to rate the impact of nausea (or vomiting) on various aspects of a patient's life (for example, ability to enjoy meals/liquids). Each item is answered using a 7 point visual analog scale with 7 being "none /not at all" and 1 being "a great deal". The two domains are summed for a total score with a possible range of 18-126. Higher scores indicate a more favorable quality of life. A total score of >108 defines those patients who had a minimal impact of Chemotherapy-Induced Nausea and Vomiting (CINV) on quality of life.
Time Frame: From (Day 2-5) to the End of Study (Day 8)
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
Number analyzed (Participants) | 34
scores on a scale | 18.3 [-76.1 to 112.8]

ADVERSE EVENTS:
Time Frame: From date of administration of study drug (Day 1) up to 192 hours (Day 8)
Arm/Group | All Participants: Palonosetron 0.25 mg/5 mL
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 3/36
Other Adverse Events (participants affected / at risk) | 13/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants: Palonosetron 0.25 mg/5 mL (N=36)
Dysphagia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants: Palonosetron 0.25 mg/5 mL (N=36)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Pyrexia (General disorders) | 2
Fatigue (General disorders) | 2
Chills (General disorders) | 1
Asthenia (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other